CLINICAL TRIAL: NCT00868530
Title: An Evaluation Of The Safety And Efficacy Of On-Demand Treatment With Xyntha (B Domain Deleted Recombinant Factor VIII, Albumin Free) In Chinese Subjects With Hemophilia A
Brief Title: Study Evaluating On-Demand Treatment Of Xyntha In Chinese Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3082B2-3316; B1831015
Record Dates: First submitted 2009-03-19; First posted 2009-03-25 (Estimated); Results first posted 2011-02-08 (Estimated); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Hemophilia A
Keywords: On-demand treatment; Hemostatic Efficacy Assessments; Factor VIII recovery; Factor VIII Inhibitor; Chinese
MeSH Terms: conditions — Hemophilia A | interventions — F8 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Xyntha (Experimental): This trial was an open-label and included assessments of safety, clinical efficacy, and Factor VIII (FVIII) recovery in Chinese subjects with hemophilia A. Subjects received on-demand treatments with Xyntha over a 6-month (calendar day) period.
  Interventions: Biological: Xyntha

INTERVENTIONS:
Biological: Xyntha — Xyntha for on-demand treatment of bleeding episodes were according to investigator prescription during the 6 months observation period. The recovery assessed by determining the Factor VIII (FVIII) concentration (FVIII:C) levels in individual subjects at the initial and final visits. The dose of Xyntha for recovery assessments is: single 50 IU/kg (±5 IU/kg) IV bolus infusion. All Xyntha administrations occurred in the clinic (hospital).

SUMMARY:
This study will evaluate the safety and efficacy of on-demand treatment with Xyntha in Chinese hemophilia A subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects equal or more than 6 years of age with mild, moderate or severe hemophilia A (FVIII activity: more than 5%, 1-5%, or less than 1%, respectively)
* Subjects with previous exposure to FVIII replacement therapy
* If human immunodeficiency virus (HIV) positive, documented cluster of differentiation (CD4) count more than 200/µL within 6 months of study entry

Exclusion Criteria:

* Diagnosed with any bleeding disorder in addition to hemophilia A
* Current FVIII inhibitor or history of FVIII inhibitor (defined as positive result of the reporting laboratory)
* Subject has no history of exposure to FVIII products (previously untreated patient [PUP])
* Subject is currently utilizing primary FVIII prophylaxis
* Subjects anticipating elective surgery that may be planned to occur in the 6 months following study entry
* Treated with immunomodulatory therapy within 30 days prior to study entry or planned use for the duration of their study participation
* Participated in another investigational drug or device study within 30 days prior to study entry or planned participation for the duration of their study participation
* Subjects with a known hypersensitivity to hamster protein
* Significant hepatic or renal impairment (alanine aminotransferase [ALT] and aspartate aminotransferase [AST] >5 x upper limit of normal [ULN], bilirubin >2 mg/dL or serum creatinine >1.25 x ULN)
* Prothrombin Time >1.5 x ULN
* Platelet count <80,000 / µL
* Pregnant or breastfeeding women
* Unwilling or unable to follow the terms of the protocol
* Any condition which may compromise the subject's ability to comply with and/or perform study-related activities or that poses a clinical contraindication to study participation, in the opinion of the Investigator or Sponsor

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2008-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- China (6):
  - Pfizer Investigational Site, Suzhou, Jiangsu
  - Pfizer Investigational Site, Heping District, Tianjin Municipality
  - Pfizer Investigational Site, Hangzhou, Zhejiang
  - Pfizer Investigational Site, Beijing
  - Pfizer Investigational Site, Guangzhou
  - Pfizer Investigational Site, Shanghai

REFERENCES:
- [Derived] Yang R, Zhao Y, Wang X, Sun J, Wu R, Jin C, Jin J, Wu D, Rendo P, Sun F, Rupon J, Huard F, Korth-Bradley JM, Xu L, Luo B, Liu YC. Safety and Efficacy of Moroctocog Alfa (AF-CC) in Chinese Patients with Hemophilia A: Results of Two Open-Label Studies. J Blood Med. 2020 Nov 25;11:439-448. doi: 10.2147/JBM.S241605. eCollection 2020. PMID 33269010
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3082B2-3316&StudyName=Study%20Evaluating%20On-Demand%20Treatment%20Of%20Xyntha%20In%20Chinese%20Subjects

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in China from September 2008 to December 2009.
Groups:
- Xyntha: Participants received on-demand treatments with Xyntha (which occurred each time a participant experienced bleeding episode during the active phase of the study) according to investigator's prescription over a 6-month (calendar day) period. A single 50 International Unit (IU)/kg (+/-5 IU/kg) intravenous (IV) bolus infusion of Xyntha was given for recovery assessments.
Period: Overall Study
Arm/Group | Xyntha
Started | 53
Completed | 49
Not Completed | 4
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Xyntha
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: Years] | 23.2 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 53

OUTCOME MEASURES:

1. Primary Outcome: Investigator Hemostatic Efficacy Assessment 8 Hours Post Infusion
Description: The Investigator Hemostatic Efficacy Assessment was based on a 4-point rating scale (Excellent = 1: definite pain relief or improvement in signs of bleeding, with no additional infusion, Good = 2: definite pain relief or improvement in signs of bleeding, Moderate = 3: probable or slight improvement, No Response = 4: no improvement at all between infusions).
Time Frame: 8 hours post infusion
Population: The Full Analysis Set (FAS) consisted of all participants who were treated and had at least 1 evaluable efficacy assessment after treatment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Xyntha
Number analyzed (Participants) | 51
Units on a scale | 1.86 (0.65)

2. Primary Outcome: Investigator Hemostatic Efficacy Assessment 24 Hours Post Infusion
Description: as for outcome 1
Time Frame: 24 hours post infusion
Population: The FAS consisted of all participants who were treated and had at least 1 evaluable efficacy assessment after treatment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Xyntha
Number analyzed (Participants) | 51
Units on a scale | 1.74 (0.61)

3. Primary Outcome: Number of Participants With Factor VIII (FVIII) Inhibitor Development
Description: Incidence of FVIII inhibitor was defined as any result determined as positive at local laboratory, and confirmed at central laboratory. Incidence was stratified by participant exposure history: Minimally Treated Patients (MTPs): those who had received at least 1 prior FVIII infusion, and <= 100 documented Exposure Days (EDs), while Previously Treated Patients (PTPs): those who had received >100 documented prior EDs. When number of prior EDs for an individual was not known to be at least 100, participants were included in the MTP population.
Time Frame: Day 1 and Month 6 or Early Termination Visit
Population: The Safety Set (SS) consisted of all participants who had taken at least 1 dose of investigational drug.
Measure: Number; unit: Participants
Arm/Group | Xyntha
Number analyzed (Participants) | 53
Participants
  MTP (n=36) | 6
  PTP (n=17) | 1

4. Secondary Outcome: FVIII Recovery : Change From Baseline in FVIII Concentration
Description: FVIII recovery was assessed by evaluating the change in FVIII concentration at 6 months compared to baseline.
Time Frame: Day 1 and Month 6 or Early Termination Visit
Population: The FAS consisted of all participants who were treated and had at least 1 evaluable efficacy assessment after treatment. Participants with missing data were not included.
Measure: Mean (Standard Deviation); unit: IU/dL per IU/kg
Arm/Group | Xyntha
Number analyzed (Participants) | 42
IU/dL per IU/kg | -0.11 (0.45)
Statistical Analysis 1: Comparison: Xyntha; Test type: Superiority or Other; p = 0.120, t-test, 2 sided

5. Secondary Outcome: Number of Participants With Less Than Expected Therapeutic Effect (LETE)
Description: The incidence of LETE, defined for on-demand treatment as no response after each of 2 successive infusions within 24 hours for the same bleeding event in the absence of confounding factors.
Time Frame: 24 hours after each of 2 successive infusion, up to 6 months
Population: The FAS consisted of all participants who were treated and had at least 1 evaluable efficacy assessment after treatment.
Measure: Number; unit: Participants
Arm/Group | Xyntha
Number analyzed (Participants) | 51
Participants | 0

6. Secondary Outcome: Number of Participants With Thrombosis Allergic-Type Reactions
Time Frame: Baseline up to 6 months
Population: The Safety Set (SS) consisted of all participants who had taken at least 1 dose of investigational drug.
Measure: Number; unit: Participants
Arm/Group | Xyntha
Number analyzed (Participants) | 53
Participants | 1

7. Secondary Outcome: Number of Participants With Thrombosis
Time Frame: Baseline up to 6 months
Population: The SS consisted of all participants who had taken at least 1 dose of investigational drug.
Measure: Number; unit: Participants
Arm/Group | Xyntha
Number analyzed (Participants) | 53
Participants | 0

8. Other Pre Specified Outcome: Frequency of Xyntha Infusions Required Per Hemorrhage
Description: The mean frequency of Xyntha infusions per hemorrhage was calculated as total number of injections throughout the study divided by total number of hemorrhagic events.
Time Frame: Day 1 to Month 6 or Early Termination Visit
Population: The FAS consisted of all participants who were treated and had at least 1 evaluable efficacy assessment after treatment.
Measure: Mean (Standard Deviation); unit: Infusions
Arm/Group | Xyntha
Number analyzed (Participants) | 51
Infusions | 1.16 (0.72)

9. Other Pre Specified Outcome: Average Dose of Xyntha Infusions Required Per Hemorrhage
Description: The average dose of Xyntha per hemorrhagic event was calculated as total dose of Xyntha throughout the study (in IU) divided by total number of hemorrhage incidence.
Time Frame: Day 1 to Month 6 or Early Termination Visit
Population: The FAS consisted of all participants who were treated and had at least 1 evaluable efficacy assessment after treatment.
Measure: Mean (Standard Deviation); unit: Dose/Bleed (IU)
Arm/Group | Xyntha
Number analyzed (Participants) | 51
Dose/Bleed (IU) | 1226.28 (1208.49)

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from the signing of the informed consent form to approximately 30 days following the Month 6/Final/Early Termination visit.
Description: Safety population = subjects who received at least 1 dose of Xyntha. The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Xyntha
Serious Adverse Events (participants affected / at risk) | 9/53
Other Adverse Events (participants affected / at risk) | 13/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Xyntha (N=53)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 1 (1)
Anti factor VIII antibody positive (Investigations) | 9 (9)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Xyntha (N=53)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 6 (8)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 1 (2)
Blood potassium decreased (Investigations) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.